CLINICAL TRIAL: NCT01003158
Title: A Phase I, Open-label, Multiple-dose, Dose-escalation Study To Assess the Safety and Tolerability of AZD8931 Monotherapy in Japanese Patients With Advanced Solid Malignancies and in Combination With Paclitaxel in Japanese Female Patients With Advanced Breast Cancer
Brief Title: Study Assessing Safety and Tolerability of AZD8931 Alone or in Combination With Paclitaxel in Japanese Patients.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0102C00010
Record Dates: First submitted 2009-10-20; First posted 2009-10-28 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Neoplasms; Metastatic Cancer; Breast Cancer
Keywords: Cancer; tumour; metastatic; breast cancer
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Breast Neoplasms | interventions — AZD 8931; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monotherapy part (Experimental): AZD8931 monotherapy
  Interventions: Drug: AZD8931
- Combination part (Experimental): AZD8931 plus paclitaxel
  Interventions: Drug: AZD8931; Drug: Paclitaxel

INTERVENTIONS:
Drug: AZD8931 — Tablet Oral bid
Drug: Paclitaxel — IV once weekly for 3 weeks followed by a week off
  Arms: Combination part

SUMMARY:
The main purpose of this study is to determine if AZD8931 can be safely administered in Japanese patients alone and in combination with weekly paclitaxel. The study will be conducted in two parts: a monotherapy and a combination part, where safe doses of study treatment will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Cancer that is refractory to standard therapies, or for which no standard therapies exist (monotherapy part)
* Patients suitable for Paclitaxel chemotherapy, who are not candidates for hormonal and anthracycline therapy (combination part)
* Life expectancy more than 12 weeks

Exclusion Criteria:

* Inadequate kidney, liver, heart, gastric, lung or eye function
* Brain metastases
* Hypersensitive to paclitaxel (combination part)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Monotherapy part: Assessment of adverse events, laboratory findings, physical examination, vital signs, ECG/UCG, chest X-ray, HRCT, SpO2 and ophthalmological examinations. | Full routine safety assessment on days 1-4, 8, 10, 14, 21, 28 then every 3 weeks after first dose of study drug
Combination part: The contents of same assessment as Monotherapy. | Full routine safety assessment on days 1-5, 8, 15, 22, 28 then every 4 weeks after first dose of study drug

SECONDARY OUTCOMES:
Combination Part: Pharmacokinetics of AZD8931 (tmax, Cmax, AUC0-10) | On Day D7 and Day D8: pre-dose then, 1, 2, 4, 6, 8 and 10 hours post dose
Combination Part: Pharmacokinetics of paclitaxel (tmax, Cmax, AUC0-10) | On Days D1 and Day D8: pre-infusion then, 0.5, 1, 1.5, 2, 4, 6, 8, 10 and 24 (D1 only) hours post start of infusion
Monotherapy Part: Pharmacokinetics of AZD8931 (Single dose plasma PK: AUC0-10, AUC0-12, AUC0-24, AUC0-t, AUC, Cmax, tmax, t1/2, CL/F, Vss/F. Multiple dose plasma PK: AUCss0-10, AUCss0-12, Cssmax, tssmax, Cssmin, CLss/F, RAC, linearity factor) | On single dose Day 1 (D1) and multiple dose Day 21 (R14): samples taken pre-dose then 1, 2, 4, 6, 8, 10, 24 (D1 only), 48 (D1 only) and 72 (D1 only) hours post dose. Day 10 (R3) and Day 14 (R7): pre-dose only

CONTACTS AND LOCATIONS:
Overall Officials: Mary Stuart, Dr., Study Director — AstraZeneca; Takayasu Kurata, Dr., Principal Investigator — Kinki University School of Medicine
Locations (1):
- Research Site, Osaka, Japan

REFERENCES:
- [Derived] Kurata T, Tsurutani J, Fujisaka Y, Okamoto W, Hayashi H, Kawakami H, Shin E, Hayashi N, Nakagawa K. Inhibition of EGFR, HER2 and HER3 signaling with AZD8931 alone and in combination with paclitaxel: phase i study in Japanese patients with advanced solid malignancies and advanced breast cancer. Invest New Drugs. 2014 Oct;32(5):946-54. doi: 10.1007/s10637-014-0112-7. Epub 2014 May 31. PMID 24875132
- See also: Reducted Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1627&filename=D0102C00010_Clinical_Study_Protocol_combined_redacted_v02a.pdf
- See also: Clinical Study Protocol Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1627&filename=AZD8931_Clinical_Study_Protocol_Redacted.pdf